CLINICAL TRIAL: NCT02974179
Title: A Long Term Follow-up Study of AMG0001 in Subjects With Critical Limb Ischemia
Status: Completed | Type: Observational
Sponsor: AnGes USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AG-CLI-0206-LTFU; 2016-003491-41 (EudraCT Number)
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Subjects who received AMG0001: Subjects from Study AG-CLI-0206 who received the study product AMG0001
  Interventions: Biological: Subjects from Study AG-CLI-0206 who received AMG0001

INTERVENTIONS:
Biological: Subjects from Study AG-CLI-0206 who received AMG0001 — Subjects from Study AG-CLI-0206 who received the study product AMG0001

SUMMARY:
Subjects from the AG-CLI-0206 phase 3 study that received AMG0001 will be eligible for the AG-CLI-0206-LTFU study

DETAILED DESCRIPTION:
The study is designed to assess the long term safety of subjects who have been treated in the phase 3 study with AMG0001. A health questionnaire will be used to collect specific information from the subject every 6 months. Only those subjects that were randomized in the AG-CLI-0206 study and who received AMG0001 are eligible to participate in this long term follow-up study. Subjects that received placebo will not be eligible for participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been treated with AMG0001 in the AG-CLI-0206 study.
* Subjects who have provided consent for this long term follow-up study either directly or through a legally authorized representative.
* Subjects who have provided a release of information to the sponsor.

Exclusion Criteria:

* Subjects who were not enrolled in the AGCLI-0206 study.
* Subjects who enrolled in AG-CLI-0206 and who were not treated with AMG0001.
* Subjects who have not provided consent to this long term follow-up study either directly or through a legally authorized representative.
* Subjects who have not provided a release of information for the Sponsor to contact them directly via phone, email and/or mail.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with critical limb ischemia who have previously been treated with AMG0001 in the AG-CLI-0206 study.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Assess the long term safety of subjects from the AG-CLI-0206 study who have been treated with AMG0001 | 3 years from the date last subject randomized into AG-CLI-0206 study
  A health questionnaire will be used to collect specific information from the subject every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Powell, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No